CLINICAL TRIAL: NCT03573180
Title: Prevalence of Dental Caries Among a Group of Egyptian Children Using Caries Assessment Spectrum and Treatment Index:A Cross Sectional Study
Brief Title: Prevalence of Dental Caries Among a Group of Egyptian Children Using CAST Index
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Aya Adel Abd El-Hafez Osman Hamza, Master student in Cairo university, Cairo University
Other Study IDs: CEBD-CU-2018-06-68
Record Dates: First submitted 2018-06-18; First posted 2018-06-29 (Actual); Last update posted 2018-06-29 (Actual); Status verified 2018-06

CONDITIONS: Dental Caries in Children
Keywords: CAST index, prevalence of caries, primary dentition caries

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to assess the prevalence of dental caries using CAST index among a group of Egyptian children in primary dentition stage.

Egyptian children aging from three to six years old attending the Outpatients' Clinic of both of Pediatric Dentistry Department, Faculty of Dentistry, Misr University for Science and Technology and the Pediatric Dentistry and Dental Public Health Department, Faculty of Dentistry, Cairo University will be examined using Caries Assessment Spectrum and Treatment

DETAILED DESCRIPTION:
* A custom made examination chart (Appendix 1) will be filled for each child including date, name, age, address, gender, medical history and any previous dental treatment. Parents' data includes: level of education and oral hygiene level.
* Prior to performing dental examination, the child will be asked to rinse his mouth with tap water and the teeth will be cleaned with cotton.
* The examiner will carefully inspect all surfaces of the teeth.
* All the primary teeth will be evaluated using CAST index as shown in Table 1.
* Each child will be given two printed sheets translated into Arabic, of his diagnosed caries status, the oral hygiene measures needed to inform the parents about the oral health status and how to keep good oral health and to indicate the need for treatment for children diagnosed with dental caries, and dietary bad habits that should be avoided to prevent caries occurrence.

Examination chart

Date:

Personal information:

Name: Age: Gender:

Address:

Medical history:

Parents' level of education:

Dental history:

Clinical examination:

E D C B A A B C D E

E D C B A A B C D E

Table 1: Caries Assessment Spectrum and Treatment(CAST) index Cast codes characteristics Code Description Concept of Health Sound 0 No visible evidence of a distinct •carious lesion is present Healthy

* Sealant 1 Pits and/or fissures are at least partially covered with a sealant material
* Restored 2 A cavity is restored with an (in)direct restorative material
* Enamel 3 Distinct visual change in enamel only. A clear caries related discoloration is visible, with or without localized enamel breakdown Reversible premorbidity
* Dentin 4 Internal caries-related discoloration in dentine. The discolored dentine is visible through enamel which may or may not exhibit a visible localized breakdown of enamel Morbidity
* 5 Distinct cavitation into dentine. The pulp chamber is intact
* Pulp 6 Involvement of the pulp chamber. Distinct cavitation reaching the pulp chamber or only root fragments are present Serious morbidity
* Abscess/ fistula 7 A pus containing swelling or a pus releasing sinus tract related to a tooth with pulpal involvement
* Lost 8 The tooth has been removed because of dental caries Mortality
* Other 9 Does not correspond to any of the other descriptions ■Severity according to CAST index:

Comments:

Dental caries: Present Absent Severity: ……………………….. (Appendix 1)

ELIGIBILITY:
Inclusion Criteria:

* Parental or guardian acceptance for participation in the study.
* Children who are medically free from any systemic diseases.
* Children with primary dentition aging from 3-6 years old.
* Both genders.

Exclusion Criteria:

* Uncooperative child.

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children will be selected from Outpatients' clinic of both of Pediatric Dentistry Department, Faculty of Dentistry, Misr University for Science and Technology and the Pediatric Dentistry and Dental Public Health Department, Faculty of Dentistry, Cairo University according to the eligibility criteria
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2018-07-01 (Estimated); Primary Completion 2018-12-31 (Estimated); Study Completion 2019-06-01 (Estimated)

PRIMARY OUTCOMES:
Prevalence of dental caries using CAST index (Frencken et al., 2013) | 6 months
  Measuring device:CAST index (Frencken et al., 2013) Measuring unit: Score (0-9)

CONTACTS AND LOCATIONS:
Overall Officials: Amr Ezzat, Professor, Study Director — Cairo University